CLINICAL TRIAL: NCT06416319
Title: Preoperative Physical Activity Improvement With the Use of Activity Trackers in Patients Undergoing Radical Cystectomy for Bladder Cancer: A Randomized Controlled Trial (PreAct)
Brief Title: Preoperative Physical Activity Improvement With the Use of Activity Trackers Before Radical Cystectomy (PreAct)
Acronym: PreAct
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Dr. Rolf M. Schwiete Foundation (Unknown)
Responsible Party: Principal Investigator, Karl-Friedrich Kowalewski, Managing Senior Physician, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-677
Record Dates: First submitted 2024-05-05; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Bladder Cancer; Bladder Neoplasm; Bladder Urothelial Carcinoma
Keywords: Cystectomy; Preoperative Exercise; Fitness Trackers; Exercise; Frailty
MeSH Terms: conditions — Urinary Bladder Neoplasms; Motor Activity; Frailty

STUDY DESIGN:
Intervention Model Description: Participants with an indication for radical cystectomy are included in this study. Recruitment, including eligibility criteria testing and randomized allocation to the intervention or control group, will take place on the day of premedication approximately 7 to 10 days prior to surgery. This period represents the prehabilitation period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Activity Goal and Feedback (Experimental): The participants in the Daily Activity Goal and Feedback arm receive a defined daily activity goal in the form of a defined number of steps, feedback on the achievement of this goal, and push-up notifications sent directly to the wristband to encourage them to remain active.
  Interventions: Device: Daily Activity Goal and Feedback
- No Daily Activity Goal or Feedback (No Intervention): The display of the fitness wristbands of the No Daily Activity Goal or Feedback arm is covered up. The participants in this arm neither receive a daily activity goal nor get feedback on the achievement of the activity goal/push-up notifications.

INTERVENTIONS:
Device: Daily Activity Goal and Feedback — The daily activity target is a fixed number of steps. The exact number of steps is determined beforehand as part of the case number planning in a pilot study with ten participants and adjusted if necessary. The activity target we suggest is 8000 steps. In addition, the participants receive feedback several times a day about the steps needed to reach the goal and whether they have ultimately reached the daily goal.
  Arms: Daily Activity Goal and Feedback

SUMMARY:
A bicentric, open-label randomised controlled trial (RCT) is planned to investigate whether the use of fitness wristbands in a defined preoperative period prior to radical cystectomy leads to a preoperative increase in participants' physical activity (number of steps per day) up to the day of radical cystectomy.

DETAILED DESCRIPTION:
The goal of the PreAct study is to test whether the use of fitness wristbands in a defined preoperative period prior to radical cystectomy with a daily activity goal and feedback on the achievement of this goal improves the participants' physical activity up to the day of radical cystectomy.

In addition to the fitness tracker, we provide each patient with a smartphone. For each fitness tracker a separate account in a fitness application is set up for (e.g. name: tracker1.0 with the corresponding e-mail address and password). Neither the patients in the Daily activity Goal and Feedback arm nor the No Daily Activity Goal or Feedback arm receive the access data to the accounts. However, the patients in the intervention group receive the access PIN for the smartphone. On this smartphone a messaging service and the fitness application are installed. The patient thus receives, for example the wristband tracker1.0, which is registered with the corresponding access data in the fitness application of the smartphone given to them. For the entire preoperative period, the Bluetooth function on the smartphone must always stay activated so that the fitness application and the fitness tracker are continuously connected to each other. A detailed description of the timing and implementation of the intervention are described in "Study design" and "Arm and Interventions".

ELIGIBILITY:
Inclusion Criteria:

* Planned radical cystectomy with bilateral pelvic lymphadenectomy and one of the different forms of urinary diversion (continent vs. incontinent; orthotopic vs. heterotopic) in patients with bladder cancer
* Participants age ≥ 18 years and capacity to consent
* Mobile participant who is not dependent on a walking aid
* The participant declares his or her consent to participate in this study by signing and dating the informed consent form prior to the surgical procedure

Exclusion Criteria:

* Karnofsky performance status scale ≤ 70% (with 70%: Care for self. Unable to carry on normal activity or to do active work (Ambulatory and capable of all selfcare but unable to carry out any work activities). ) (Range: 0 - 100 percent with 0 percent "participant´s death" and 100 percent "no disabilities"
* ASA Physical Status Classification: ASA > 3 (3: A patient with severe systemic disease)
* ASA 1, 2, 3 if acute or chronic diseases of the musculoskeletal system or the central nervous system are involved that result in a symptomatic restriction of motor and / or, in the last case, neurological function (healing ruptures and fractures, Parkinson's disease, multiple sclerosis, etc.)
* Emergency intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Number of steps per day | Participants' daily step count is recorded on the day of surgery when the fitness tracker is put down.
  Average daily step count measured by the fitness tracker during the period of prehabilitation 7 to 10 days before surgery.

SECONDARY OUTCOMES:
Total number of steps | Participants' total number of steps is recorded on the day of surgery when the fitness tracker is put down.
  Total number of steps measured by the fitness tracker during the period of prehabilitation 7 to 10 days before surgery.
Postoperative physical activity | Morning of postoperative day 4 at 7 PM
  The postoperative physical activity of the participants measured by the average number of steps per day and in total on postoperative days 1 to 3. Neither arm will receive a daily activity goal. However, the fitness trackers of the No Daily Activity Goal or Feedback arm are still covered.
Postoperative Complications | On postoperative day 30 and 90
  Postoperative complications measured by the Comprehensive Classification Index (CCI), on a scale from 0 (no complications) to 100 (death), (Slankamenac, Graf et al. 2013) and the Clavien-Dindo Classification (CDC), which consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V), the first one indicating any deviation from the normal postoperative course, the highest grade indicating death (Clavien, Barkun et al. 2009):
  CDC ≥ 3a corresponding to a CCI ≥ 26.2 defined as "severe complications" including CDC = 5 and CCI = 100 defined as "patient's death" and the total number of complications
Operating time | On the day of surgery
  In minutes, incision - surgical incision closure
Blod loss | On the day of surgery
  In millilitres
Required transfusion of blood products | On the day of surgery
  Number of red blood cell concentrates, platelet concentrates, frozen fresh plasma
Feasibility of the planned urinary diversion | On the day of surgery
  Yes or no
Conversion rate | On the day of surgery
  If the planned urinary diversion is not feasible
Patient Reported Outcome Measures (PROMs) | On the day of randomization at the premedication appointment and on the day of discharge which is on average 2 weeks after the surgery and postoperative day 30 and 90
  SF-36: Health-related quality of life (Scale 0 - 100: The higher the score, the lower the disability. A score of 100 corresponds to no disability)
Length of hospital stay (LOS) | On the day of discharge which is on average 2 weeks after the surgery
  LOS measured by the number of days spent in the hospital after surgery until discharge
Readmission rate | On postoperative day 90 if occured
  Readmissions due to a complication of the radical cystectomy
Reoperation rate | On postoperative day 90 if occured
  Reoperation due to a complication of the radical cystectomy
Length of stay in the intensive care unit (ICU) | On postoperative day 90 if occured
  Days spent in the ICU after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Friedrich Kowalewski, PD Dr. med, Principal Investigator — Department of Urology, University Medical Center Mannheim, Heidelberg University
Locations (2):
- Germany (2):
  - Department of Urology, University Medical Center Mannheim, University of Heidelberg, Mannheim, Baden-Wurttemberg
  - Urologische Klinik München Planegg (UKMP), München, Bavaria